CLINICAL TRIAL: NCT03436212
Title: Real-Life Home Glucose Monitoring Over 14 Days in T2D Patients With Intensified Therapy Using Insulin Pump. The CLOSE Study
Brief Title: Real-Life Home Glucose Monitoring Over 14 Days in T2D Patients With Intensified Therapy Using Insulin Pump.
Acronym: CLOSE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Air Liquide Santé International (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: ALMED-17-001
Record Dates: First submitted 2018-02-12; First posted 2018-02-19 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Continuous Glucose Monitoring

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Continuous Glucose Monitoring (CGM) (Other): DEXCOMG4 device for 14 days
  Interventions: Device: Continuous Glucose Monitoring (CGM)

INTERVENTIONS:
Device: Continuous Glucose Monitoring (CGM) — DEXCOMG4 device

SUMMARY:
This study aims at describing the glucose level by automated glucose sensors and correlating it with insulin delivery and meals over 14 days in insulin-requiring T2D patients living in real-life conditions.

ELIGIBILITY:
Selection criteria:

* Type 2 Diabetes diagnosed for at least 5 years
* Treated with insulin pump for at least 6 months
* 7.5% ≤ HBA1c ≤ 10% (last available value dated less than 3 months)
* Having given his/her free, express and informed consent to participate to the study

Inclusion Criteria:

* 7.5% ≤ HBA1c ≤ 10% (result of the dosage performed at selection visit)
* Daily insulin requirement ≤ 1.5U/kg/day
* Having been compliant to take pictures of his/her meals and snacks over the 3 days prior to the inclusion visit

Non-selection/Non-inclusion criteria:

* Pregnant or breastfeeding woman
* Comorbidity which, in the investigator's opinion, could jeopardize the study completion
* Patient with difficulties to understand the study procedures or deemed unfit, by the Investigator, to comply with operating instructions of CGM equipment.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2017-09-05 (Actual); Primary Completion 2018-03-06 (Actual); Study Completion 2018-03-06 (Actual)

PRIMARY OUTCOMES:
Relationships between glucose levels and insulin doses | 14 days
  To describe the relationships between glucose levels and insulin doses between meals and at meal-times in T2D patients using pumps over 14 days.

CONTACTS AND LOCATIONS:
Overall Officials: Yves Reznik, MD, Study Chair — CHU CAEN
Locations (1):
- CHU de Caen, Service Endocrinologie, Diabétologie, Caen, France